CLINICAL TRIAL: NCT07310836
Title: A Retrospective Study of Safety and Efficacy of Locoregional Therapies Combined With Anti-VEGF/TKIs and Immune Checkpoint Inhibitors for All Comers of Intention-to-treat Patients With Hepatocellular Carcinoma Beyond UCSF Criteria Before Liver Transplantation
Status: Not yet recruiting | Type: Observational
Sponsor: Ningbo Medical Center Lihuili Hospital (Other Government)
Responsible Party: Principal Investigator, lucaide, Chief Physician/Professor, Ningbo Medical Center Lihuili Hospital
Other Study IDs: KY2025PJ483
Record Dates: First submitted 2025-12-16; First posted 2025-12-30 (Actual); Last update posted 2025-12-30 (Actual); Status verified 2025-12

CONDITIONS: Hepatocellular Carcinoma; Liver Transplantation
MeSH Terms: conditions — Carcinoma, Hepatocellular

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Beyond UCSF Criteria Cohort: HCC patients receiving conversion therapy beyond UCSF criteria
  Interventions: Combination Product: Locoregional Therapy (LRT) + Systemic Drug Therapy
- Within UCSF Criteria Cohort: HCC patients within UCSF Criteria Cohort

INTERVENTIONS:
Combination Product: Locoregional Therapy (LRT) + Systemic Drug Therapy — Treatment regimens, doses, and durations varied based on individual clinical decisions and are collected retrospectively.
  Groups: Beyond UCSF Criteria Cohort

SUMMARY:
This is a single-center, retrospective cohort study aiming to evaluate the safety and efficacy of a combined treatment strategy for patients with hepatocellular carcinoma (HCC) who are beyond the UCSF criteria but intended for liver transplantation. The primary objective is to assess the outcomes of these "intention-to-treat" patients who received locoregional therapies (LRT, such as TACE or radiotherapy) in combination with systemic therapy (anti-VEGF/Tyrosine Kinase Inhibitors and Immune Checkpoint Inhibitors) as a "conversion therapy" prior to potential transplantation. This approach is distinct from traditional bridging or down-staging therapies by incorporating more aggressive systemic regimens. The study plans to enroll 300 subjects. The exposure group will include approximately 100 patients beyond UCSF criteria who received the combined conversion therapy between January 2020 and December 2024. A control group of about 200 patients who met the UCSF criteria and were directly listed for transplantation in the same period will be used for comparison. Data will be collected from medical records and the China Liver Transplant Registry (CLTR), with follow-up until December 2025.

Primary outcome measures include:

Objective Response Rate (ORR) of conversion therapy per mRECIST. Rate of successful down-staging to meet UCSF criteria.

1-, 2-, and 3-year overall survival (OS) rates of the intention-to-treat population.

Actual liver transplantation rate after successful conversion. Post-transplant 1-, 2-, and 3-year OS and recurrence-free survival (RFS) rates.

Secondary outcomes involve:

Safety profiles of both conversion therapy and subsequent transplantation. Analysis of factors influencing conversion success and treatment efficacy. Determination of an optimal washout period for Immune Checkpoint Inhibitors prior to transplantation.

The study seeks to provide high-level evidence for optimizing pre-transplant conversion strategies for advanced HCC patients currently outside standard transplant criteria.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥16;
* Clinical diagnosis of HCC;
* CNLC Stage I-IIIA.

Exclusion Criteria:

* Extrahepatic metastasis;
* Type IV portal vein tumor thrombus.

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: This retrospective, single-center cohort study plans to include 300 patients with HCC. All patients were managed at the study center between January 1, 2020, and December 31, 2024.
  1. Beyond UCSF Criteria Cohort (n = 100): Patients with HCC tumors exceeding the UCSF transplant criteria but intended for liver transplantation. All patients in this cohort received multimodal conversion therapy, combining locoregional therapies with systemic therapy.
  2. Within UCSF Criteria Cohort (n = 200): A control group of patients whose HCC tumors met the UCSF criteria at the time of listing and were directly registered for liver transplantation without receiving the aforementioned conversion therapy.
Sampling Method: Non-Probability Sample
Enrollment: 300 (Estimated)
Dates: Start 2025-12-20 (Estimated); Primary Completion 2025-12-31 (Estimated); Study Completion 2026-03-31 (Estimated)

PRIMARY OUTCOMES:
Objective Response Rate (ORR) | From the start of conversion therapy until the completion of therapy (assessed up to 24 months).
  Proportion of patients achieving a Complete Response (CR) or Partial Response (PR) according to mRECIST criteria during the conversion therapy period.
Successful Down-staging Rate to UCSF Criteria | From the start of conversion therapy until the date of meeting UCSF criteria or therapy termination (assessed up to 24 months).
  Proportion of patients whose tumor burden is reduced to meet the UCSF transplant criteria after conversion therapy, based on imaging and tumor marker assessment.
1/2/3-year Overall Survival (OS) Rate | From the initiation of conversion therapy, assessed at 1, 2, and 3 years.
  The proportion of patients who received conversion therapy and are still alive at 1, 2, and 3 years after the transplantation surgery, analyzed using the Kaplan-Meier method.

CONTACTS AND LOCATIONS:
Overall Officials: Caide Lu, Professor, Principal Investigator — Ningbo Medical Centre Lihuili Hospital

IPD SHARING:
Plan to Share IPD: Undecided
A specific plan for sharing de-identified individual participant data (IPD) from this retrospective study is under development. The final decision will depend on several factors, including but not limited to: institutional review board (IRB) approval, compliance with data privacy regulations, and the establishment of appropriate data use agreements. If shared, the data would likely include demographic, clinical treatment, tumor response, and survival outcome data to support validation of study findings. The research team is committed to evaluating the possibility of sharing data in a manner that protects participant confidentiality and contributes to scientific knowledge.